CLINICAL TRIAL: NCT05002543
Title: CORCYM Mitral, Aortic aNd Tricuspid Post-maRket Study in a reAl-world Setting
Acronym: MANTRA
Status: Recruiting | Type: Observational
Sponsor: Corcym S.r.l (Industry)
Responsible Party: Sponsor
Other Study IDs: LNH800
Record Dates: First submitted 2021-07-26; First posted 2021-08-12 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Cardiac Valve Disease
Keywords: Aortic Valve Replacement; Mitral Valve Replacement; Mitral Valve Repair; Tricuspid Valve Repair
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- MANTRA Aortic Sub-study: Subjects diagnosed with aortic valve disease who are considered suitable to undergo aortic valve replacement with a CORCYM device can be included in this study.
  The following devices can be entered in the study:
  Tissue Valve:
  * Perceval® PLUS SUTURELESS AORTIC HEART VALVE
  * Perceval® S SUTURELESS AORTIC HEART VALVE
  Mechanical Valves:
  * Bicarbon™ Bileaflet Heart Valve Prostheses Models:
    * Bicarbon Fitline Aortic (LFA)
    * Bicarbon Slimline Aortic (LSA)
    * Bicarbon Overline Aortic (LOV)
  * Carbomedics Prosthetic Heart Valve Models:
    * Standard Aortic Valve
    * Reduced Aortic Valve
    * Supra-Annular Aortic Valve (Top Hat)
    * Orbis™ Aortic Valve
  Ascending Aorta Prostheses
  * CARBOMEDICS-CARBO-SEAL™
  * CARBOMEDICS CARBO-SEAL™ VALSALVA
- MANTRA Mitral/Tricuspid Sub-study: Subjects diagnosed with mitral and/or tricuspid valve disease who are considered suitable to undergo mitral valve repair/replacement and/or tricuspid valve repair with a CORCYM device can be included in this study.
  The following devices can be entered in the study:
  Annuloplasty Rings:
  * SOVERING™ ANNULOPLASTY DEVICE models
    * annuloplasty ring, mitral model
    * annuloplasty band, mitral and tricuspid models
  * Carbomedics Annuloplasty Ring models:
    * CARBOMEDICS ANNULOFLO®
    * CARBOMEDICS ANNULOFLEX®
  * Memo Annuloplasty Ring o MEMO 3D™ SEMIRIGID ANNULOPLASTY RING
  Mitral Valves:
  * Bicarbon™ Bileaflet Heart Valve Prostheses Models:
    o Bicarbon Fitline Mitral (LFM)
  * Carbomedics Prosthetic Heart Valve Models:
    * Standard Mitral Valve
    * Orbis™ Mitral Valve
    * OptiForm® Mitral Valve
- MANTRA Memo 4D Sub-study: Subjects diagnosed with mitral valve disease who are considered suitable to undergo mitral valve repair with a CORCYM Memo 4D annuloplasty ring can be included in this study.

SUMMARY:
MANTRA is a prospective, multiple-arm, multi-center, global, post-market clinical follow-up study. The main objective is to monitor ongoing safety and performance of the CORCYM devices and accessories used for aortic, mitral and tricuspid valvular diseases in a real-world setting.

Corcym S.r.l., is a medical device manufacturer with a broad product portfolio for cardiac surgeons, offering solutions for the treatment of aortic, mitral and tricuspid valve disease.

The MANTRA Master Plan (Master Protocol) is intended as an overarching Umbrella Protocol that allows multiple sub-studies to be added, as needed. The Umbrella Master Protocol concept offers an excellent solution to provide post-marketing clinical follow-up information on the entire cardiac surgery heart valve portfolio of the sponsor in a common database, including corelab assessment of hemodynamic and structural performance, annular motion and Dynamics for one of the products.

Currently, three sub-studies are planned:

* MANTRA - Aortic Sub-Study
* MANTRA - Mitral/Tricuspid Sub-Study (Excluding Memo 4D)
* MANTRA - Memo 4D Sub-Study

DETAILED DESCRIPTION:
The MANTRA Master Plan (Master Protocol) is intended as an overarching Umbrella Protocol that allows multiple substudies to be added, as needed. The Umbrella Master Protocol concept offers an excellent solution to provide post-marketing clinical follow-up information on the entire cardiac surgery heart valve portfolio of the sponsor in a common database.

Currently, three substudies are planned:

* MANTRA - Aortic Sub-Study
* MANTRA - Mitral/Tricuspid Sub-Study (excluding Memo 4D)
* MANTRA - Memo 4D Sub-Study

The aim of the studies assembled under the master protocol is the continued collection of safety and performance data during heart valve procedures and the relevant follow-up visits in subjects where any of the CORCYM devices and accessories are used in a real-world setting, in accordance with the IFUs, and at the discretion of the investigator.

MANTRA study is expected to enroll approximately 2150 subjects in up to 130 sites worldwide:

* Approximately 1650 subjects considered suitable for treatment with a CORCYM aortic device
* Approximately 300 subjects considered suitable for treatment with a CORCYM mitral and/or tricuspid device (excluding Memo 4D)
* Approximately 200 subjects considered suitable for treatment with Memo 4D

Expected enrollment duration may vary across the different projects. Subject follow-up is planned at discharge, 30 days after implantation and then annually up to 10 years. Sites can choose to participate in one or more sub-studies.

All available data shall be gathered during standard medical care.

At a minimum, the following data will be collected:

* Informed Consent
* Screening/Baseline data, including demographics and medical history
* Procedural data
* Hospitalization and Discharge data
* Follow-up data: 30 days and annually up to 10 years post procedure
* Serious Adverse Event and Device Deficiencies information

As part of the study, the subject will be asked to complete quality of life questionnaire(s) at baseline, 30 days and at 1-year follow-up.

In addition, for the MEMO 4D sub-study only, an Echocardiography Core Laboratory has been appointed by the Sponsor to assess the hemodynamic and structural performance, annular motion and dynamics, and 3D echocardiogram images (transesophageal during the procedure and transthoracic during follow up) will be collected for Corelab readings.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated approved Informed Consent
* Subject is willing and able to comply with the follow up schedule of the protocol
* Eligible for treatment with CORCYM aortic, mitral and/or tricuspid products as outlined in the applicable Instructions for Use (IFU)

Exclusion Criteria:

* Subject is already participating to another clinical investigation that could confound the results of this clinical investigation.
* Subject has a life expectancy ≤ 12 months
* Subject has contraindications to the use of CORCYM aortic, mitral and/or tricuspid devices as outlined in the applicable Instructions For Use (IFU)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects diagnosed with heart valve disease who are considered suitable to undergo heart valve replacement/repair with a CORCYM device can be included
Sampling Method: Probability Sample
Enrollment: 2150 (Estimated)
Dates: Start 2021-06-29 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint in the AORTIC Sub-study is number and percentage of subjects with Device Success | 30 days
  Device success at 30 days (+14 days) based on VARC-3, defined as:
  * Technical success
  * Freedom from mortality
  * Freedom from surgery or intervention related to the device or to a major vascular or access-related or cardiac structural complication
  * Intended performance of the valve (mean gradient<20 mmHg and less than moderate aortic regurgitation)
  The number and percentage of subjects with device success at 30 days as per VARC-3 definition, along with individual component of the success, will be presented.
The primary endpoint in the MITRAL/TRICUSPID Sub-study is number and percentage of subjects with Device Success | 30 days
  Device success at 30 days (+14 days) based on MVARC, defined as:
  * Procedural mortality or stroke AND
  * Proper placement and positioning of the device AND
  * Freedom from unplanned surgical or interventional procedures related to the device or access procedure AND
  * Continued intended safety and performance of the device, including:
    * Evidence of structural or functional failure
    * Specific device-related technical failure issues and complications
    * MITRAL: Reduction of Mitral Regurgitation (MR) to either optimal or acceptable levels (site-reported)
    * TRICUSPID: Reduction of Tricuspid Regurgitation (TR) to either optimal or acceptable levels (site-reported)
  Number and percentage of subjects with device success, along with individual component, will be presented.
The primary endpoint in the MEMO 4D Sub-study is number and percentage of subjects with Device Success | 30 days
  Device success at 30 days (+14 days) based on the MVARC, defined as:
  * Procedural mortality or stroke; AND
  * Proper placement and positioning of the device; AND
  * Freedom from unplanned surgical or interventional procedures related to the device or access procedure; AND
  * Continued intended safety and performance of the device, including:
    * Evidence of structural or functional failure
    * Specific device-related technical failure issues and complications
    * Reduction of Mitral Regurgitation (MR) to either optimal or acceptable levels without significant mitral stenosis (i.e., post-procedure EOA is ≥ 1.5 cm2 with a transmitral gradient <5 mmHg), and with no greater than mild MR core-lab assessed
  The number and percentage of subjects with device success at 30 days as per MVARC definition, along with individual component of the success, will be presented.

SECONDARY OUTCOMES:
Mortality (all-cause mortality, cardiovascular mortality, device related mortality) | up to 10 years from implant
  Number of patients with this event
Major Adverse Cardiovascular and Cerebrovascular Event (MACCE - composite endpoint of all cause death, myocardial infarction, stroke, and valve re-intervention) | up to 10 years from implant
  Number of patients with this event
Re-hospitalization (all-cause re-hospitalization, cardiovascular re-hospitalization, device related re-hospitalization) | up to 10 years from implant
  Number of patients with this event
Technical success | intraoperatively
  Technical success, defined as successful delivery, correct positioning and deployment of the first intended device intraoperatively
Clinical Efficacy (AORTIC sub-study) | 12 months
  Clinical Efficacy according to VARC-3 guidelines
Valve-related long-term clinical efficacy | at 5 years and up to 10 years
  Valve-related long-term clinical according to VARC-3 guidelines
Bioprosthetic Valve Dysfunction (BVD), including Structural Valve Deterioration (SVD), Non structural valve dysfunction (NSVD), Thrombosis and Endocarditis | up to 10 years from implant
  Number of patients with this event
Patient outcome (Kansas City Cardiomyopathy Questionnaire (KCCQ-12); and EQ-5D-5L (in patients treated with Perceval Plus) | 12 months
  Quality of life improvement from baseline up to 12 months
Patient outcome (New York Heart Association (NYHA) Classification) | up to 10 years from implant
  Change of New York Heart Association (NYHA) functional class from baseline up to 12 months after implant, and at each subsequent follow-up
Hemodynamic and structural performance | up to 10 years from implant
  Main hemodynamic parameters will be collected according to the different indications (Aortic, Mitral and Tricuspid)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Gaggianesi, Study Director — Corcym S.r.l
Locations (52):
- United States (9):
  - St. Vincent Heart Center of Indiana, Indianapolis, Indiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - Duke University, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - University Hospitals Cleveland, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Lankenau Institute for Medical Research, Wynnewood, Pennsylvania
- Innsbruck Medical University, Innsbruck, Austria
- Belgium (3):
  - Ziekenhuis Oost Limburg, Genk
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
- Canada (3):
  - University of Calgary (Foothills Hospital), Calgary
  - Hospital Laval IUCPQ, Québec
  - St. Michael's Hospital, Toronto
- France (4):
  - CHU Clermont-Ferrand_Hopital Gabriel Montpied, Clermont-Ferrand
  - Centre Hospitalier de Lens, Lens
  - CHU Poitiers, Poitiers
  - CHU Toulouse_Rangueil University Hospital, Toulouse
- Germany (8):
  - Universitätsklinikum Augsburg, Augsburg
  - Kerckhoff Klinik, Bad Nauheim
  - Deutsches Herzzentrum Berlin, Berlin
  - Herzzentrum Dresden Universitätsklinik, Dresden
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Magdeburg, Magdeburg
  - Klinikum Nürnberg, Nuremberg
  - Klinikum Oldenburg GGMBH AöR, Oldenburg
- Italy (12):
  - Ospedale Riuniti Ancona, Ancona
  - Policlinico S.Orsola-Malpighi, Bologna
  - Fondazione Poliambulanza Istituto Ospedaliero, Brescia
  - Ospedale Città di Lecce, Lecce
  - Ospedale del Cuore "G. Pasquinucci", Massa
  - IRCCS Policlinico San Donato, Milan
  - Azienda ospedaliera dei Colli - Ospedale Monaldi, Napoli
  - Policlinico Paolo Giaccone, Palermo
  - A.O.U. Citta della Salute e della Scienza di Torino - Ospedale Molinette, Torino
  - Ospedale Cà Foncello di Treviso, Treviso
  - Az. Ospedaliero-Universitaria "Ospedali Riuniti" di Trieste, Trieste
  - Ospedale San Bortolo, Vicenza
- Netherlands (2):
  - Catharina Ziekenhuis, Eindhoven
  - UMC Groningen, Groningen
- Hospital de Santa Maria Lisbon, Lisbon, Portugal
- Dedinje Cardiovascular Institute, Belgrade, Serbia
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Yonsei University Severance Cardiovascular Hospital, Seoul
  - Pusan National University Yangsan Hospital, Yangsan
- Switzerland (2):
  - Inselspital, Universitätsspital Bern, Bern
  - Stadtspital Triemli, Zurich
- United Kingdom (3):
  - Queen Elisabeth Medical Centre, Birmingham
  - Bristol Royal Infirmary, Bristol
  - King's College Hospital, London

REFERENCES:
- [Derived] Dzemali O, Rodriguez Cetina Biefer H, Di Eusanio M, Fabre O, Troise G, Bonaros N, Grimaldi F, Choi YH, Santarpino G, Baeza C, Pollari F, Marcheix B, Pacini D, Argano V, Baghai M, Bhabra M, Mazzaro E, Badano L, Kempfert J. Mitral valve repair with the semi-rigid Memo 4D annuloplasty ring: early clinical and echocardiographic outcomes from the MANTRA study. Interdiscip Cardiovasc Thorac Surg. 2024 Dec 25;40(1):ivae208. doi: 10.1093/icvts/ivae208. PMID 39666948
- [Derived] Micovic S, Nobre A, Choi JW, Solinas M, Shehada SE, Torella M, Baeza C, Parrino E, Pollari F, Troise G, Kappert U, Mellert F, Je HG, Argano V, Lam KY, Rinaldi M, Gutermann H, Meuris B; MANTRA Investigators. Early outcomes of aortic valve replacement with Perceval PLUS sutureless valve: results of the prospective multicentric MANTRA study. J Cardiothorac Surg. 2024 Jun 21;19(1):340. doi: 10.1186/s13019-024-02861-1. PMID 38902742